CLINICAL TRIAL: NCT00359021
Title: An Open-label Trial With TMC125 as Part of an ART Including TMC114/Rtv and an Investigator-selected OBR in HIV-1 Infected Subjects Who Participated in a DUET Phase III Trial (TMC125-C206 or TMC125-C216).
Brief Title: An Open-label Trial With TMC125 in Patients Who Have Virologically Failed in a DUET Trial (TMC125-C206 or TMC125-C216).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002740; TMC125-C217 (Other: Tibotec Pharmaceuticals); TMC125-C206 (Other: Tibotec Pharmaceuticals); TMC125-C216 (Other: Tibotec Pharmaceuticals)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: HIV-1
Keywords: HIV-1; treatment experienced; virologic failure
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): TMC125 200 mg twice daily until commercially available
  Interventions: Drug: TMC125

INTERVENTIONS:
Drug: TMC125 — 200 mg twice daily until commercially available

SUMMARY:
The purpose of this trial is to evaluate the long-term safety and tolerability of TMC125 200 mg twice daily as part of an antiretroviral therapy including TMC114/rtv and an investigator selected optimized background in HIV-1 infected patients who have participated in a DUET trial (TMC125-C206 or TMC125 C216) and have met the definition of virologic failure at Week 24 or later in these trials.

DETAILED DESCRIPTION:
This is a Phase III open-label, roll-over trial to evaluate the long term tolerability, safety, antiviral and immunological effect of TMC125 as part of an individually optimized antiretroviral therapy including TMC114/rtv in HIV-1 infected patients who participated in one of the DUET (TMC125-C206 or TMC125-C216) trials. Also the change in HIV-1 resistance over time will be evaluated. This trial offers patients meeting the definition of virologic failure at Week 24 or beyond the option to roll-over to an open-label trial where they will receive TMC125 and TMC114/rtv. Three hundred patients are estimated to enroll into this trial. The withdrawal visit of the DUET trial will be the first visit of this trial. From this visit onward, all patients will receive 200 mg twice daily TMC125 and 600/100 mg twice daily TMC114/rtv until both TMC114 and TMC125 are commercially available or the therapy is no longer of clinical benefit to the patient. Patients will receive an antiretroviral therapy consisting of TMC125 as the only non-nucleoside reverse transcriptase inhibitor (NNRTI), TMC114/rtv as the only protease inhibitor (PI) and an optimized background, which will be selected by the investigator according to the local standard of care, the patient's experience with previous therapies and most recent resistance testing. The most recent HIV-1 genotype-analysis system report results from the DUET trial will be made available. TMC125 will be dosed at 200 mg twice daily, administered orally as 2 tablets twice daily with food.TMC114/rtv will be dosed at 600/100 mg twice daily, administered orally as 2 tablets TMC114 and 1 capsule ritonavir twice daily with food.The optimized background will comprise of at least 1 approved ARV drug: 1 or more NRTI(s), with or without ENF. Administration will continue until both TMC114 and TMC125 are commercially available or therapy is no longer of clinical benefit to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient was previously randomized in a DUET (TMC125-C206 or TMC125-C216) trial and completed at least 24 weeks of treatment
* Patient was virologically failing in a DUET trial.

Exclusion Criteria:

* Use of disallowed concomitant therapy
* Any grade 4 toxicity according to the Division of AIDS (DAIDS) grading table
* Patients who had to be withdrawn from the DUET (TMC125-C206 or TMC125-C216) trials because of any of the mandatory withdrawal criteria of that trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2006-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (72):
- United States (32):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Springs, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Fort Laudersale, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Camden, New Jersey
  - Newark, New Jersey
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
  - Seattle, Washington
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Neuquén
  - San Juan Bautista
- Darlinghurst, Australia
- Belgium (2):
  - Antwerp
  - Liège
- Brazil (4):
  - Curitiba
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Canada (4):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
  - Toronto
- Chile (2):
  - Providencia
  - Santiago
- France (9):
  - Bordeaux
  - Le Kremlin-Bicêtre
  - Lyon
  - Marseille
  - Paris
  - Rennes
  - Toulouse
  - Tourcoing
  - Villejuif
- Germany (5):
  - Berlin
  - Essen
  - Hamburg
  - Mannheim
  - München
- Mexico (2):
  - Mex Ctity
  - Mexico City
- Panama City, Panama
- San Juan, Puerto Rico
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- Thailand (2):
  - Bangkok
  - Khon Kaen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with human immunodeficiency virus - type 1 (HIV-1) infection were enrolled in this study from DUET Study TMC125-C206 or TMC125-C216 and met the definition of virologic failure at Week 24 or later in these studies, or who completed one of the DUET studies after 96 weeks of treatment.
Groups:
- DUET PLACEBO: Participants who received Placebo in a previous DUET study and received open-label treatment with 200 mg twice daily etravirine, also known as TMC125 (ETR) and 600/100 mg twice daily darunavir (DRV)/low-dose ritonavir (rtv) were referred to as ETR-naïve participants.
- DUET TMC125: Participants who received etravirine, also known as TMC125 (ETR) in a previous DUET study and received open-label treatment with 200 mg twice daily ETR and 600/100 mg twice daily darunavir (DRV)/low-dose ritonavir (rtv) were referred to as ETR-experienced participants.
Period: Overall Study
Arm/Group | DUET PLACEBO | DUET TMC125
Started | 256 | 247
Completed | 175 | 195
Not Completed | 81 | 52
Not completed — Adverse Event | 26 | 8
Not completed — Subject Non-Compliant | 1 | 2
Not completed — Subject Ineligible To Continue The Trial | 1 | 0
Not completed — Subject Reached A Virologic Endpoint | 45 | 32
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 4 | 1
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DUET PLACEBO | DUET TMC125 | Total
Number analyzed (Participants) | 256 | 247 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 245 | 497
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.28) | 46.6 (7.01) | 46.7 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 37 | 64
  Male | 229 | 210 | 439

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Adverse Events
Description: The table below provides the number of participants who experienced Serious Adverse Events (SAEs) and Other Adverse Events (except SAEs) that started or worsened in severity during the overall TMC125-C217 treatment period. The duration of treatment ranged per patient from 1 week to 180 weeks, with a median of 62 weeks.
Time Frame: 1 week to 180 weeks, with a median of 62 weeks
Population: The safety analysis was carried out on the ITT population, which included all participants who received at least one dose of investigational medication.
Measure: Number; unit: Participants
Groups:
- DUET PLACEBO: Participants who received Placebo in a previous DUET study received open-label treatment with 200 mg twice daily etravirine, also known as TMC125 (ETR) and 600/100 mg twice daily darunavir (DRV)/low-dose ritonavir (rtv) were referred to as ETR-naïve participants.
- All Participants: DUET Placebo + DUET TMC125
Arm/Group | DUET PLACEBO | DUET TMC125 | All Participants
Number analyzed (Participants) | 256 | 247 | 503
Participants
  Serious Adverse Events (SAEs) | 46 | 42 | 88
  Other Adverse Events (AEs) | 160 | 137 | 297

2. Secondary Outcome: The Percentage of Participants With Virologic Outcomes Over Time
Description: The table below shows the percentage of participants with virologic suppression (< 50 copies/mL), the percentage of participants who were virologic failures (VF) (>50 copies/mL, discontinued prior to time X for reasons of VF or for other reasons, except for VF or adverse event, with a last viral load >50 copies/mL), and the percentage of participants with no viral load (VL) data available over time (ie, at Weeks 24, 48, and 96).
Time Frame: Weeks 24, 48, and 96
Population: The intent-to-treat (ITT) population was used as the primary analysis population for the efficacy analysis and included all participants who took at least one dose of etravirine (ETR) (also known as TMC125) in the TMC125-C217 study.
Measure: Number; unit: Percentage of Participants
Arm/Group | DUET PLACEBO | DUET TMC125
Number analyzed (Participants) | 256 | 247
Percentage of Participants
  Week 24 - Virologic Response (<50 cop/mL) | 43.0 | 62.3
  Week 24 - Virologic Failure | 46.9 | 31.6
  Week 24 - No VL Data available | 10.2 | 6.1
  Week 48 - Virologic Response (<50 cop/mL) | 35.2 | 44.5
  Week 48 - Virologic Failure | 50.4 | 31.2
  Week 48 - No VL Data available | 14.5 | 24.3
  Week 96 -Virologic Response (<50 cop/mL) | 7.4 | 4.5
  Week 96 - Virologic Failure | 48.0 | 27.5
  Week 96 - No VL Data available | 44.5 | 68.0

3. Secondary Outcome: Change in Plasma Viral Load Versus Baseline (ie, Mean Change in log10 Plasma Viral Load From Baseline Over Time)
Description: In the table below, the total number of participants analyzed in the Duet Placebo and Duet TMC125 groups, respectively at each time point were: Baseline (256;247 participants), Week 24 (251;240 participants), Week 48 (235;192 participants), and Week 96 (123;69 participants).
Time Frame: Baseline, Week 24, Week 48, and Week 96
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | DUET PLACEBO | DUET TMC125
Number analyzed (Participants) | 256 | 247
log10 copies/mL
  Week 24 | -0.8 [-0.93 to -0.63] | 0 [-0.11 to 0.03]
  Week 48 | -0.7 [-0.86 to -0.54] | -0.1 [-0.16 to -0.02]
  Week 96 | -0.5 [-0.66 to -0.30] | -0.2 [-0.38 to -0.04]

ADVERSE EVENTS:
Time Frame: 07-Jun-2006 to 24-Jan-2012.
Description: All "Serious Adverse Events (SAEs)" emerging during the TMC125-C217 treatment period are reported below; "Other Adverse Events (not including SAEs)" provided below occurred in at least 0.5% of participants. The duration of the TMC125 treatment period ranged per patient from 1 week to 180 weeks, with a median of 62 weeks.
Groups:
- All Participants: Participants who received placebo or TMC125 in a previous DUET study (DUET Placebo + DUET TMC125).
Arm/Group | DUET PLACEBO | DUET TMC125 | All Participants
Serious Adverse Events (participants affected / at risk) | 46/256 | 42/247 | 88/503
Other Adverse Events (participants affected / at risk) | 160/256 | 137/247 | 297/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DUET PLACEBO (N=256) | DUET TMC125 (N=247) | All Participants (N=503)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2 | 4
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0 | 3
Cerebral toxoplasmosis (Infections and infestations) | 1 | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Cryptococcosis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 1 | 2
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus myelomeningoradiculitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 2 | 4
HIV infection (Infections and infestations) | 0 | 1 | 1
Hepatitis c (Infections and infestations) | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Histoplasmosis (Infections and infestations) | 1 | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 1 | 0 | 1
Keratitis fungal (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Papilloma viral infection (Infections and infestations) | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 3 | 0 | 3
Pneumonia (Infections and infestations) | 5 | 4 | 9
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Pyomyositis (Infections and infestations) | 1 | 0 | 1
Pyothorax (Infections and infestations) | 1 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 2 | 2 | 4
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1
Strongyloidiasis (Infections and infestations) | 1 | 0 | 1
Tuberculosis of central nervous system (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arteriogram coronary (Investigations) | 1 | 0 | 1
Blood amylase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Female reproductive tract carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Coma (Nervous system disorders) | 0 | 1 | 1
Dementia (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 3
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 0 | 1 | 1
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 1
Breast cosmetic surgery (Surgical and medical procedures) | 1 | 0 | 1
Liposuction (Surgical and medical procedures) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DUET PLACEBO (N=256) | DUET TMC125 (N=247) | All Participants (N=503)
Diarrhoea (Gastrointestinal disorders) | 32 | 24 | 56
Nausea (Gastrointestinal disorders) | 20 | 15 | 35
Injection site nodule (General disorders) | 14 | 8 | 22
Pyrexia (General disorders) | 13 | 6 | 19
Bronchitis (Infections and infestations) | 18 | 12 | 30
Herpes simplex (Infections and infestations) | 32 | 17 | 49
Influenza (Infections and infestations) | 18 | 18 | 36
Nasopharyngitis (Infections and infestations) | 21 | 15 | 36
Oral candidiasis (Infections and infestations) | 23 | 14 | 37
Sinusitis (Infections and infestations) | 19 | 23 | 42
Upper respiratory tract infection (Infections and infestations) | 14 | 11 | 25
Urinary tract infection (Infections and infestations) | 14 | 8 | 22
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 | 15 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 14 | 21
Headache (Nervous system disorders) | 18 | 10 | 28
Insomnia (Psychiatric disorders) | 13 | 7 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 26
Rash (Skin and subcutaneous tissue disorders) | 24 | 4 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees that before he/she publishes any results of this trial, he/she shall provide the sponsor with at least 45 days for full review of the pre-publication manuscript prior to submission of the manuscript to the publisher.